CLINICAL TRIAL: NCT06080373
Title: Formulation-Based Cognitive-Behavioral Therapy Compared to an Active Control and a Waitlist in Adult Inmates With ADHD: A Randomized Controlled Trial
Brief Title: Formulation-based CBT for Adult Inmates With ADHD: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Valencia (Other)
Responsible Party: Principal Investigator, Carlos López-Pinar, Proffesor, Universidad Europea de Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UEuropeaValencia
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Formulated-based cognitive behavioral therapy (Experimental): Participants randomized to the CBT group will receive a minimum of 13 and a maximum of 22 sessions of individual formulation-based CBT. It will be delivered by psychologists trained in CBT, according to a manual that will be available soon. Prior to intervention, a behavioral assessment is conducted to operationalize each case's clinically relevant behaviors, antecedents, and maintenance stimuli. Each case will be formulated and presented to the participant in simple and easy to understand language. To illustrate this, a schematic formulation of the typical case of an adult with ADHD is shown in Figure 2. Specific behavioral goals will then be agreed upon for each participant. To achieve these goals, various treatment strategies will be presented in the following sessions. The choice of strategies, the order in which they are applied, and the duration of each module will be customized for each participant according to the case formulation.
  Interventions: Behavioral: Formulation-based cognitive behavioral therapy
- PROBECO and social therapeutic establishments (Active Comparator): The Spanish participants assigned to the active control group will receive the PROBECO. It is a group program designed by the Spanish Penitentiary Agency for its application with inmates convicted of different types of violent crimes . Its main goals are to eradicate criminal behavior and reduce recidivism, to modify the relevant dynamic risk factors related to general delinquency, and to introduce new social skills and prosocial values. It consists of four phases: (I) general intervention: aimed at the acquisition of social skills; (II) specific intervention: consists of four specific educational itineraries; (III) relapse prevention; (IV) follow-up.
  Similarly, German participants will be assigned to a special type of prison known as a social therapeutic facility, where they will undergo compulsory psychotherapy focused primarily on relapse prevention.
  Interventions: Behavioral: PROBECO
- Waitlist (No Intervention): Participants in waitlist control group will receive no treatment while experimental groups are treated. They will be offered to receive CBT after the study.

INTERVENTIONS:
Behavioral: PROBECO — Spanish participants in the active control group will undergo the PROBECO program, designed by the Spanish Penitentiary Agency for various violent crimes. It aims to eradicate criminal behavior, reduce recidivism, and teach social skills. It has four phases.
  German participants will be placed in social therapeutic facilities for compulsory psychotherapy focused on relapse prevention.
  Arms: PROBECO and social therapeutic establishments
Behavioral: Formulation-based cognitive behavioral therapy — The CBT program includes these core modules:
  A. ADHD Psychoeducation: Provides information on ADHD characteristics, neurobiology, treatments, and their efficacy. Shared with a significant other if available.
  B. Planning Skills and Distraction Management: Teaches time management, task prioritization, and distraction control techniques.
  C. Cognitive Restructuring: Based on Ellis' Rational Behavioral Emotive Therapy, it helps participants identify and modify irrational thoughts for better emotional regulation.
  D. Maintenance of Treatment Gains: Reviews progress, identifies risk factors, and develops action plans for post-treatment challenges.
  Arms: Formulated-based cognitive behavioral therapy

SUMMARY:
Background Recent literature suggests that ADHD is a risk factor for the development of antisocial behavior that is more severe and persistent than in community and other psychiatric populations. The combination of stimulant medication and psychotherapy (particularly cognitive-behavioral therapy, CBT) is considered an evidence-based intervention for adults with ADHD. In contrast, few studies have evaluated the efficacy of medication in adult prisoners with ADHD, and the literature on the efficacy of psychotherapy is virtually nonexistent. Therefore, this article presents the protocol of a trial that will assess the efficacy of a formulation-based CBT program for inmates with ADHD.

Methods The study has a multicenter randomized controlled trial design. After screening and recruitment, participants will be randomly assigned to the CBT intervention, a general offender treatment program, or a waitlist. Pre- and post-treatment self-report and clinician-report assessments, as well as 6- and 12-month follow-up assessments will be conducted. These will include both clinical (e.g., ADHD symptoms, depression and anxiety symptoms, self-esteem, alcohol/drug abuse, treatment adherence, quality of life) and criminological (e.g., recidivism and risk of recidivism) measures. Linear mixed models will be used to assess differences between groups.

Discussion This study may be the first to evaluate the efficacy of a psychotherapy intervention in adult inmates with ADHD. It is expected that addressing the specific needs of ADHD would not only result in the previously reported clinical improvements (e.g., reduction in ADHD and comorbidity symptoms), but also reduce the risk and rate of recidivism compared to the general intervention or no intervention. However, the design may be limited by the difficulties inherent in the prison setting and in following up the sample after release.

ELIGIBILITY:
Inclusion Criteria:

* To have signed written informed consent to participate in the study
* To be between 18 and 65 years of age
* To meet the DSM-5 diagnostic criteria for ADHD (American Psychiatric Association, 2013)
* To have been convicted of at least one crime under Spanish or German criminal law
* To have been incarcerated for at least six months and three or fewer years since the completion of the conviction at the time of eligibility assessment.

Exclusion Criteria:

* To have a severe personality disorder, psychotic disorder, or pervasive developmental disorder as their primary diagnosis, as the intervention would not meet their clinical needs
* To have an IQ of 80 or less, as measured by a standardized IQ test (Raven et al., 1993), due to the complexity of the cognitive components in the CBT program
* To have participated in a previous psychological intervention for ADHD;
* To not be fluent in Spanish or German, depending on the study site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Conners Adult ADHD Diagnostic Interview for DSM-IV (CAADID) | Pre and post-treatment plus follow-up assessments 6 and 12 months after the end of the intervention
  This is considered one of the primary outcomes. The CAADID is a structured interview divided into two parts. Part I may be self-administered or clinician-administered and collects information on the subject's demographic history, developmental history, associated risk factors, and comorbidity, while Part II must be administered by a trained clinician and assesses DSM-IV criteria for ADHD in adults. Only Part II will be used for the study, as information on patient history is not relevant for measuring response to interventions.
Reoffending rate | Pre and post-treatment plus follow-up assessments 6 and 12 months after the end of the intervention
  This will be the primary criminological outcome. Police records will be checked every 6 months after the end of treatment to look for new arrests. We will also try to check court and prison records for new convictions and incarcerations. However, access to this information may be very limited in European criminal justice systems, so it may be difficult to obtain.

SECONDARY OUTCOMES:
Clinical Global Impression (CGI) | Pre and post-treatment plus follow-up assessments 6 and 12 months after the end of the intervention
  Is a three-item observer-rated scale that measures illness severity, global improvement or change, and therapeutic response. It is a widely used, robust measure of efficacy in clinical trials. The global functioning outcome provides a measure of the impact that symptoms have on daily functioning in life domains (e.g., social, family, work, personal, and academic, among others).
Attention-deficit/hyperactivity rating scale-IV | Pre and post-treatment plus follow-up assessments 6 and 12 months after the end of the intervention
  This measure will be the primary self-reported outcome. The scale includes 18 items that reference DSM-IV criteria (American Psychiatric Association, 2000), and it is used to determine the presence and severity of current ADHD symptoms. Each item is scored from 0 (never, rarely) to 3 (often). This measure has high validity and reliability and has been widely used both for clinical and research purposes.
Rosenberg self-esteem scale (RSES | Pre and post-treatment plus follow-up assessments 6 and 12 months after the end of the intervention
  This 10-item scale provides a unidimensional measure of global self-esteem and acceptance of self-worth.
Adult ADHD Quality of Life Questionnaire (AAQoL | Pre and post-treatment plus follow-up assessments 6 and 12 months after the end of the intervention
  It is an ecologically valid measure of the quality of life designed specifically for adults with ADHD. It consists of 29 items corresponding to four domains particularly relevant for patients with ADHD: productivity, psychological health, social relationships, and life perspectives.
Maudsley Addiction Profile (MAP) | Pre and post-treatment plus follow-up assessments 6 and 12 months after the end of the intervention
  This is a 60-item, multidimensional instrument for assessing treatment outcome in people with drug and/or alcohol problems.
Beck depression inventory-II (BDI-II) and Beck anxiety inventory (BAI) | Pre and post-treatment plus follow-up assessments 6 and 12 months after the end of the intervention
  These are one of the most commonly used self-report instruments to assess the severity of depressive and anxiety symptoms, respectively. A total score is obtained from the sumo of its 21 items, with higher scores indicating higher levels of depression or anxiety.
Historical Clinical Risk Management-20 (HCR-20) | Pre and post-treatment plus follow-up assessments 6 and 12 months after the end of the intervention
  This instrument is a guide to predicting violence risk in inmates and psychiatric patients, providing a probabilistic prediction of the risk of future antisocial behavior. A trained rater must assess the presence of 20 past, present, and future risk factors organized into three different scales. The HCR-20 includes both dynamic and static risk factors. Three levels of risk can be identified without initial reference to explicit tables, scales, or cutoff points: low, moderate, or high (and imminent).

OTHER OUTCOMES:
Treatment adherence | During the intervention
  In order to measure adherence more objectively, attendance at treatment sessions and completion of homework assignments are systematically recorded by the therapist at each session.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos López-Pinar, Dr, Principal Investigator — Universidad Europea de Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopez-Pinar C, Martinez-Sanchis S, Carbonell-Vaya E, Martinez-Raga J, Retz W. Formulation-based cognitive behavioral therapy compared to an active control and a waitlist in adult inmates with ADHD: study protocol for a randomized controlled trial. Trials. 2024 Sep 6;25(1):594. doi: 10.1186/s13063-024-08434-w. PMID 39243058